CLINICAL TRIAL: NCT01280487
Title: A Phase 1b, Multi-Center, Open Label, Uncontrolled, Serial Cohort, Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Daily Oral Doses of ZSTK474 in Subjects With Advanced Solid Malignancies
Brief Title: A Safety Study of Oral ZSTK474 in Patients With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zenyaku Kogyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSTK474-101
Record Dates: First submitted 2011-01-18; First posted 2011-01-20 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Neoplasms
Keywords: ZSTK474; PI3K inhibitor
MeSH Terms: conditions — Neoplasms | interventions — ZSTK474

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral ZSTK474 (Experimental): Daily oral dosing for 21 days per cycle
  Interventions: Drug: ZSTK474

INTERVENTIONS:
Drug: ZSTK474 — Daily oral dosing for 21 days each cycle

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and preliminary efficacy of daily oral doses of ZSTK474, an oral phosphatidylinositol 3-kinase (PI3K) inhibitor, in subjects with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females ≥18 years of age;
2. Histologically-confirmed advanced (metastatic or unresectable) solid tumor - for which available therapy is not effective;
3. ECOG performance status score of ≤2 and an expected survival of >8 weeks;
4. Recovered from the toxicities of prior chemotherapy, radiotherapy, and other cancer therapies; all toxicities must be determined to be below Grade 2 (assessed using the NCI CTCAE v4.0).
5. Adequate blood counts with a hemoglobin (Hgb) of ≥9.0 mg/dL, absolute neutrophil count (ANC) >1,500/mm3, and platelets ≥100,000/mm3 (all without transfusion support);
6. Subjects who are willing and able to provide written informed consent.

In the expanded cohort at the MTD only: Subjects must be willing to undergo mandatory biopsies of tumor tissue twice during the first cycle (before and during dosing) and must have tumor tissue in a location accessible to incisional biopsy of a superficial lesion or percutaneous core needle biopsy on an outpatient basis without undue risk to the subject.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding;
2. Men or women of reproductive potential who are not willing to use acceptable means of contraception while on study drug and for an additional 90 days after the last dose of study drug;
3. Body Mass Index (BMI) is ≥30 kg/m2;
4. Have primary central nervous system (CNS) tumors or untreated/uncontrolled CNS metastases; Note: Subjects with stable/controlled CNS metastases may be enrolled (i.e., if CNS lesions have been stable in size for at least one month and the subject is off steroid and anti-convulsants).
5. Have received any investigational interventional agents within the 4 weeks prior to the start of dosing with ZSTK474;
6. Are receiving concurrent anti-tumor chemotherapy, radiotherapy, or immunotherapy - or have received any of these non-investigational agents within the previous 4 weeks or 5-half-lives (whichever is longer) prior to the start of dosing with ZSTK474;
7. Are not able or willing to comply with the study procedures, including the study visit schedule;
8. Have previously been treated with a phosphatidylinositol 3 kinase (PI3K) inhibitor;
9. Have serious or significant intercurrent illnesses or underlying diseases, such as:

   1. Diabetes
   2. Gastrointestinal disorder
   3. Hepatic: AST or ALT >2.5 x ULN (or >5.0 x ULN with liver metastases) or serum bilirubin >1.5 x ULN;
   4. Renal (acute or chronic renal disease or eGFR <55 mL/min)
   5. Cardiovascular:

      * Uncontrolled hypertension or blood pressure >140/90 mmHg;
      * Symptomatic congestive heart failure;
      * Myocardial infarction within the past 6 months;
      * Unstable angina pectoris;
      * Cardiac arrhythmia;
      * Congenital long QT syndrome;
      * QTc >450 msec for men or >470 msec for women.
   6. Other:

      * Known diagnosis of HIV infection;
      * Other ongoing or active infections;
      * Psychiatric illness, substance abuse or social situation that would preclude study compliance.
      * Other serious concurrent illness that would preclude assessment of drug effect;
      * PT/PTT)/APTT/INR >ULN for subjects not on anti-coagulants; INR > 1.5 x ULN for subjects on low dose warfarin.
10. Current treatment with the following drugs:

    * any anti-seizure medications;
    * therapeutic anti-coagulant doses of warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 21 days

SECONDARY OUTCOMES:
Pharmacokinetics | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Craig Lockhart, MD, Principal Investigator — Washington University School of Medicine; Anthony Olszanski, MD, Principal Investigator — Fox Chase Cancer Center; Geoffrey Shapiro, MD PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania